CLINICAL TRIAL: NCT00599586
Title: Randomized Controlled Trial of Treating Migraine With Acupuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Liang Fanrong, Acupuncture & Tuina college of chengdu univeristy of TCM
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006CB5045011; 2006CB5045011 (Other Grant/Funding Number: 973 program)
Record Dates: First submitted 2008-01-03; First posted 2008-01-24 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Migraine
Keywords: migraine; acupuncture; efficacy; safety; meridian; acupoint
MeSH Terms: conditions — Migraine Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- group 1 (Experimental): specific acupoints of Shaoyang meridians
  Interventions: Other: acupuncture
- Group 2 (Experimental): Non-specific acupoints of Shaoyang meridians
  Interventions: Other: acupuncture
- group 3 (Experimental): Acupoints of other meridians
  Interventions: Other: acupuncture
- group 4 (Sham Comparator): Non-acupoints
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — Subjects are treated five days a week continuously, and for four weeks.They are treated 30min every time.
  Other Names: electro-acupuncture

SUMMARY:
The purpose of the study is to testify whether acupuncture is effective for migraine, and provide evidence for the hypothesis that"Acupuncture effect is based on meridians, and gathering of meridian Qi is the key point."

DETAILED DESCRIPTION:
The purpose of the study is to testify whether acupuncture is effective for migraine, through treating migraine patients for a month, using different acupoints according to literatures of treating migraine with acupuncture, and try to provide clinical evidence for the hypothesis that"Acupuncture effect is based on meridians, and gathering of meridian Qi is the key point."

ELIGIBILITY:
Inclusion Criteria:

1. Age of a subject is older than 18 and is younger than 65.(The subject is younger than 50 when he was ill for the first time.)
2. Consistent with the diagnostic criteria of Premonitory Migraine and Non- Premonitory Migraine.
3. Attacks of migraine are equal to or more than 2 times in the last three months.
4. With more than one year history of migraine
5. Informed consent is signed by a subject or his lineal relation.

Exclusion Criteria:

1. With serious protopathy or disease of cardiovascular, liver, renal,gastrointestinal, hematological systems and so on.
2. Psychotic，patients with allergic constitution or easily getting infected or bleeding.
3. Patients have used drugs for preventing migraine in the last four weeks.
4. Pregnant women or women in lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
number of days with migraine | 4 weeks
frequency of migraine attacks | 4 weeks

SECONDARY OUTCOMES:
Migraine-Specific Quality-of-Life Questionnaire | a month
Transcranial Doppler Sonography | a month

CONTACTS AND LOCATIONS:
Overall Officials: Fan-rong Liang, master, Study Chair — Chengdu University of TCM
Locations (1):
- Chengdu University of TCM, Chengdu, Sichuan, China

REFERENCES:
- [Result] Linde K, Streng A, Jurgens S, Hoppe A, Brinkhaus B, Witt C, Wagenpfeil S, Pfaffenrath V, Hammes MG, Weidenhammer W, Willich SN, Melchart D. Acupuncture for patients with migraine: a randomized controlled trial. JAMA. 2005 May 4;293(17):2118-25. doi: 10.1001/jama.293.17.2118. PMID 15870415
- [Derived] Zheng H, Huang W, Li J, Zheng Q, Li Y, Chang X, Sun G, Liang F. Association of pre- and post-treatment expectations with improvements after acupuncture in patients with migraine. Acupunct Med. 2015 Apr;33(2):121-8. doi: 10.1136/acupmed-2014-010679. Epub 2014 Dec 30. PMID 25549933
- [Derived] Deng ZQ, Zheng H, Zhao L, Zhou SY, Li Y, Liang FR. Health economic evaluation of acupuncture along meridians for treating migraine in China: results from a randomized controlled trial. BMC Complement Altern Med. 2012 Jun 14;12:75. doi: 10.1186/1472-6882-12-75. PMID 22697367
- [Derived] Li Y, Zheng H, Witt CM, Roll S, Yu SG, Yan J, Sun GJ, Zhao L, Huang WJ, Chang XR, Zhang HX, Wang DJ, Lan L, Zou R, Liang FR. Acupuncture for migraine prophylaxis: a randomized controlled trial. CMAJ. 2012 Mar 6;184(4):401-10. doi: 10.1503/cmaj.110551. Epub 2012 Jan 9. PMID 22231691
- [Derived] Zhao L, Zhang FW, Li Y, Wu X, Zheng H, Cheng LH, Liang FR. Adverse events associated with acupuncture: three multicentre randomized controlled trials of 1968 cases in China. Trials. 2011 Mar 24;12:87. doi: 10.1186/1745-6215-12-87. PMID 21435214
- [Derived] Li Y, Liang F, Yu S, Liu X, Tang Y, Yang X, Tian X, Yan J, Sun G, Chang X, Zheng H, Zhang H, Ma T. Randomized controlled trial to treat migraine with acupuncture: design and protocol. Trials. 2008 Oct 20;9:57. doi: 10.1186/1745-6215-9-57. PMID 18928574